CLINICAL TRIAL: NCT02353026
Title: A Phase I Study of Intravenous Artesunate in Patients With Solid Tumors
Brief Title: Phase I Study of Intravenous Artesunate for Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro028
Record Dates: First submitted 2015-01-27; First posted 2015-02-02 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous Artesunate (Experimental): Intravenous Artesunate administered on Day 1 and 8 every 3 weeks
  Interventions: Drug: Intravenous Artesunate

INTERVENTIONS:
Drug: Intravenous Artesunate — Intravenous Artesunate in escalating doses: 8, 12, 18, 25, 34, 45 mg/kg on days 1 and 8 of every 3 week cycles

SUMMARY:
This is a Phase One study to determine the safety, tolerability, and maximum tolerated dose of intravenous artesunate in patients with solid tumors. A rapid dose escalation design will be used, in which single patients will be enrolled to escalating dose levels until a grade 2 or higher toxicity occurs during cycle 1. Enrollment will then continue using 3 to 6 patients at each dose level until a dose is reached at which 2 or more patients out of 6 experience a treatment-related toxicity.

DETAILED DESCRIPTION:
A rapid dose escalation design will be used, in which single patients will be enrolled to each dose level until a grade >/= 2 treatment-related toxicity occurs during cycle 1; enrollment then will proceed using a classic 3+ 3 dose escalation design. If the toxicity was grade 2, then enrollment will continue on that dose level. If the toxicity was grade 3 or 4, then enrollment will continue on one dose level below that dose. Dose escalation with the 3+3 design will continue until >/= 2 patients out of 6 experience a treatment-related dose-limiting toxicity. Then, the maximum tolerated dose and recommended Phase II dose of intravenous artesunate will be one dose level below the level at which the toxicities occurred.

ELIGIBILITY:
Inclusion Criteria:

* At least one measurable lesion by RECIST criteria
* Willing to undergo pharmacogenetic testing
* Over the age of 18 years and able to provide informed consent
* No standard of care therapy available which has a proven overall survival benefit
* Adequate kidney, liver, and bone marrow function
* Life expectancy of greater than 3 months
* ECOG performance status less than or equal to 2

Exclusion Criteria:

* Chemotherapy or surgery within 4 weeks of treatment start
* Radiation treatment within 3 weeks prior to treatment start
* Untreated brain metastases or neurologically unstable CNS metastases
* Any severe or uncontrolled medical condition or other condition which could affect participation in the study including: unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction </= 6 months prior to study entry
* Previous diagnosis of alpha- or beta-thalassemia
* Patients on a medication or herbal therapy known to inhibit CYP2A6, UGT1A9, or UGT2B7
* Female patients who are pregnant or breast feeding, or adult patients who are of reproductive potential and are unwilling to refrain from conceiving a child during study treatment
* Patients unwilling or unable to comply with the protocol, or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 1 year
  One dose level below the dose at which 2 or more out of 6 patients experienced dose-limiting toxicities

CONTACTS AND LOCATIONS:
Overall Officials: John F Deeken, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Deeken JF, Wang H, Hartley M, Cheema AK, Smaglo B, Hwang JJ, He AR, Weiner LM, Marshall JL, Giaccone G, Liu S, Luecht J, Spiegel JY, Pishvaian MJ. A phase I study of intravenous artesunate in patients with advanced solid tumor malignancies. Cancer Chemother Pharmacol. 2018 Mar;81(3):587-596. doi: 10.1007/s00280-018-3533-8. Epub 2018 Feb 1. PMID 29392450